CLINICAL TRIAL: NCT01165216
Title: Phase 1 Study of Ipilimumab (BMS-734016) in Combination With Paclitaxel and Carboplatin in Japanese Patients With Non-Small Cell Lung Cancer
Brief Title: Japanese Study of Ipilimumab Administered in Combination With Paclitaxel/Carboplatin in Patients With Nonsmall-cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA184-113
Record Dates: First submitted 2010-07-16; First posted 2010-07-19 (Estimated); Results first posted 2014-07-22 (Estimated); Last update posted 2014-07-22 (Estimated); Status verified 2014-06

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Ipilimumab; Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dose Level 1: Ipilimumab, 3 mg/kg + Paclitaxel + Carboplatin (Experimental): Participants received ipilimumab, 3 mg/kg, administered as a single dose intravenously (IV) over 90 minutes every 3 weeks, plus paclitaxel, 175 mg/m^2 , administered as a single dose IV over 3 hours every 3 weeks (up to 6 doses), and carboplatin, area under the curve (AUC)=6, administered as a single dose IV over 30-60 minutes every 3 weeks (up to 6 doses).
  Interventions: Drug: Ipilimumab, 3 mg; Drug: Paclitaxel; Drug: Carboplatin
- Dose Level 2: Ipilimumab, 10 mg/kg + Paclitaxel + Carboplatin (Experimental): Participants received ipilimumab, 10 mg/kg, administered as a single dose IV over 90 minutes every 3 weeks, plus paclitaxel, 175 mg/m^2 , administered as a single dose IV over 3 hours every 3 weeks (up to 6 doses), and carboplatin, AUC=6, administered as a single dose IV over 30-60 minutes every 3 weeks (up to 6 doses).
  Interventions: Drug: Ipilimumab, 10 mg; Drug: Paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Drug: Ipilimumab, 3 mg — Intervenous (IV) injection, administered every 3 weeks for up to 6 cycles
  Arms: Dose Level 1: Ipilimumab, 3 mg/kg + Paclitaxel + Carboplatin
Drug: Ipilimumab, 10 mg — IV injection, administered every 3 weeks for up to 6 cycles
  Other Names: BMS-734016
  Arms: Dose Level 2: Ipilimumab, 10 mg/kg + Paclitaxel + Carboplatin
Drug: Paclitaxel — IV injection, 175 mg/m^2, administered every 3 weeks for up to 6 cycles
Drug: Carboplatin — IV injection, AUC=6, administered every 3 weeks for up to 6 cycles. (AUC=area under the concentration curve)

SUMMARY:
The primary purpose of this study was to establish the recommended dose of ipilimumab administered in combination with paclitaxel and carboplatin in Japanese patients with nonsmall-cell lung cancer.

ELIGIBILITY:
Key Inclusion Criteria:

* Histologically or cytologically documented nonsmall-cell lung cancer (NSCLC) presenting as stage IIIB disease without indications for definitive radiotherapy, stage IV disease, or recurrent disease following radiation therapy or surgical resection
* No prior chemotherapy, hormonal therapy, immunotherapy, or targeted-therapy-containing regimens for the treatment of NSCLC
* Life expectancy of at least 3 months
* Eastern Cooperative Oncology Group performance score of 0-1
* Adequate bone marrow function
* Hemoglobin ≥9.0 g/dL
* Absolute neutrophil count ≥1,500/mm^3
* Platelet count ≥100,000/mm^3
* Adequate liver function
* Total bilirubin level ≤2.0*the upper limit of normal (ULN)
* Asparate aminotransferase level ≤2.5*ULN
* Alanine aminotransferase level ≤2.5*ULN
* Adequate renal function
* Calculated creatinine clearance based on Cockcroft and Gault formula ≥50 mL/min.

Key Exclusion Criteria:

* Symptomatic central nervous system (CNS) metastasis or active CNS metastasis requiring medication
* Malignant body cavity fluid (eg, pleural effusion, cardiac effusion, ascites) that recurred despite appropriate supportive care
* Prior radiation of ≥30% of major bone-marrow containing areas (pelvis, lumbar spine)
* Documented history of severe autoimmune or immune-mediated symptomatic disease that required prolonged (longer than 2 months) systemic immunosuppressant treatment
* Documented history of motor neuropathy considered of autoimmune origin (eg, Guillain Barré syndrome)
* Any concurrent malignancy other than nonmelanoma skin cancer, carcinoma in situ of the cervix, carcinoma in situ of the breast, carcinoma of the mucous membrane of the gastrointestinal tract, or superficial bladder cancer treated with systemic therapy
* ≥Grade 2 diarrhea
* History of or concurrent disease of gastrointestinal tract perforations
* ≥Grade 2 peripheral neuropathy (motor or sensory)
* Uncontrolled intercurrent illness including infection requiring systemic therapy, symptomatic congestive heart failure, uncontrolled hypertension, uncontrolled angina pectoris, uncontrolled peptic ulcer, and cardiac arrhythmia requiring medication
* Positive finding for human immunodeficiency virus antibody, hepatitis B surface antigen, or hepatitis C virus antibody.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2010-09; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Chuo-ku, Tokyo, Japan

REFERENCES:
- [Derived] Horinouchi H, Yamamoto N, Fujiwara Y, Sekine I, Nokihara H, Kubota K, Kanda S, Yagishita S, Wakui H, Kitazono S, Mizugaki H, Tokudome T, Tamura T. Phase I study of ipilimumab in phased combination with paclitaxel and carboplatin in Japanese patients with non-small-cell lung cancer. Invest New Drugs. 2015 Aug;33(4):881-9. doi: 10.1007/s10637-015-0243-5. Epub 2015 May 1. PMID 25924991
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were enrolled in successive cohorts of 3 to 6 patients, using a standard 3+3 design. Of 15 patients enrolled, all received some treatment (chemotherapy or ipilimumab); 12 received at least 1 dose of ipilimumab.
Groups:
- Dose Level 1: Ipilimumab, 3 mg/kg + Paclitaxel + Carboplatin: Participants received ipilimumab, 3 mg/kg, administered as a single dose intravenously (IV) over 90 minutes every 3 weeks, plus paclitaxel, 175 mg/m^2 , administered as a single dose IV over 3 hours every 3 weeks (up to 6 doses), and carboplatin, area under the concentration curve (AUC)=6, administered as a single dose IV over 30-60 minutes every 3 weeks (up to 6 doses).
- Dose Level 2: Ipilimumab, 10 mg/kg + Paclitaxel + Carboplatin: Participants received ipilimumab, 10 mg/kg, administered as a single dose IV over 90 minutes every 3 weeks, plus paclitaxel, 175 mg/m^2, administered as a single dose IV over 3 hours every 3 weeks (up to 6 doses), and carboplatin, AUC=6, administered as a single dose IV over 30-60 minutes every 3 weeks (up to 6 doses).
Period: Overall Study
Arm/Group | Dose Level 1: Ipilimumab, 3 mg/kg + Paclitaxel + Carboplatin | Dose Level 2: Ipilimumab, 10 mg/kg + Paclitaxel + Carboplatin
Started | 8 (Participants who received any study drug) | 7 (Participants who received any study drug)
Received at Least 1 Dose of Ipilimumab | 6 | 6
Completed | 0 (Completed=still on study drug) | 0 (Completed=still on study drug)
Not Completed | 8 | 7
Not completed — Adverse Event | 6 | 3
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Disease progression | 1 | 3

BASELINE CHARACTERISTICS:
Population: All participants who received at least 1 dose of study drug.
Groups:
- Dose Level 1: Ipilimumab, 3 mg/kg + Paclitaxel + Carboplatin: Participants received ipilimumab, 3 mg/kg, administered as a single dose intravenously (IV) over 90 minutes every 3 weeks, plus paclitaxel, 175 mg/m^2, administered as a single dose IV over 3 hours every 3 weeks (up to 6 doses), and carboplatin, area under the concentration curve (AUC)=6, administered as a single dose IV over 30-60 minutes every 3 weeks (up to 6 doses).
- Total: Total of all reporting groups
Arm/Group | Dose Level 1: Ipilimumab, 3 mg/kg + Paclitaxel + Carboplatin | Dose Level 2: Ipilimumab, 10 mg/kg + Paclitaxel + Carboplatin | Total
Number analyzed (Participants) | 8 | 7 | 15
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.0 (12.62) | 58.9 (10.25) | 57.3 (11.26)
Age, Customized [Number; unit: Participants]
  Younger than 65 years | 7 | 4 | 11
  65 years and older | 1 | 3 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 6 | 6 | 12
Race/Ethnicity, Customized [Number; unit: Participants]
  Japanese | 8 | 7 | 15
  Not reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing a Dose-limiting Toxicity (DLT)
Description: A DLT was defined as study drug-related adverse event occurring during the first 2 cycles after ipilimumab administration in the induction phase and was any of the following: Grade 4 absolute neutrophil count (ANC) decreased (<500 cells/ mm^3) for 7 or more consecutive days; febrile Neutropenia (body temperature ≥38.5° C with ANC <1000 /mm^3) lasting >3 days; Grade 4 platelet count decreased (<25,000 cells/mm^3) or Grade 3 platelet count decreased requiring a platelet transfusion; Grade 3 or greater nausea, vomiting, diarrhea, despite the use of adequate/maximal medical intervention; Grade 3 or greater aspartate transaminase/alanine transaminase level and rash that has not resolved to Grade 2 or lower within 2 weeks after onset; or any Grade 3 or greater nonhematologic toxicity (except Grade 3 fatigue, Grade 3 asthenia, Grade 3 transient arthralgia/myalgia, or Grade 3 transient abnormal electrolyte levels).
Time Frame: Day 1 of Cycles 1 and 2 From Day 1 of Cycle 3 to Day 21 of Cycle 4
Population: Participants who received at least 1 dose of ipilimumab
Measure: Number; unit: Participants
Groups:
- Dose Level 2: Ipilimumab, 10 mg/kg + Paclitaxel + Carboplatin: Participants received ipilimumab, 10 mg/kg, administered as a single dose IV over 90 minutes every 3 weeks, plus paclitaxel, 175 mg/m^2, administered as a single dose IV over 3 hours every 3 weeks (up to 6 doses) and carboplatin, AUC=6, administered as a single dose IV over 30-60 minutes every 3 weeks (up to 6 doses).
Arm/Group | Dose Level 1: Ipilimumab, 3 mg/kg + Paclitaxel + Carboplatin | Dose Level 2: Ipilimumab, 10 mg/kg + Paclitaxel + Carboplatin
Number analyzed (Participants) | 6 | 6
Participants | 2 | 1

2. Secondary Outcome: Number of Participants With Death As Outcome, Serious Adverse Events (SAEs), Drug-related SAEs, Drug-related Adverse Events (AEs), AEs Leading to Discontinuation, Drug-related AEs Leading to Discontinuation
Description: AE=any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that may not have a causal relationship with treatment. SAE=a medical event that at any dose results in death, persistent or significant disability/incapacity, or drug dependency/abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization. Treatment-related=having certain, probable, possible, or unknown relationship to study drug. AE incidence was assessed from Day 1 until Week 24 and every 12 weeks thereafter during the maintenance period, until discontinuation of study drug, due to progression of disease, toxicities requiring discontinuation, withdrawal of consent, or study closure, and at least every 4 weeks(±1 week) until all study drug-related toxicities had recovered to resolved, stabilized or returned to baseline or were deemed irreversible during the follow-up period).
Time Frame: Continuously from Day 1 to Week 24 and every12 weeks thereafter during maintenance until discontinuation of drug
Population: Participants who received at least 1 dose of any study drug
Measure: Number; unit: Participants
Arm/Group | Dose Level 1: Ipilimumab, 3 mg/kg + Paclitaxel + Carboplatin | Dose Level 2: Ipilimumab, 10 mg/kg + Paclitaxel + Carboplatin
Number analyzed (Participants) | 8 | 7
Participants
  Deaths | 0 | 0
  SAEs | 3 | 1
  Drug-related SAEs | 3 | 1
  Drug-related AEs | 8 | 7
  AEs leading to discontinuation | 6 | 3
  Drug-related AEs leading to discontinuation | 6 | 3

3. Secondary Outcome: Number of Participants With Best Overall Response (BOR) of Partial Response (PR) or Stable Disease
Description: Tumor response was determined for all participants with measurable lesions by radiologic responses as defined by Response Evaluation Criteria in Solid Tumors (RECIST), version 1.1. The BOR was the best response recorded from start of treatment until disease progression/recurrence. RECIST for target lesions: PR=at least a 30% decrease in the sum of the longest dimension (LD) of target lesions, taking as reference the baseline sum LD; stable disease=neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease, taking as reference the smallest sum LD since the treatment started. At minimum, tumor measurements were to be obtained at screening, every 6 weeks (±1 week) during the induction phase and every 12 weeks (±1 week) during the maintenance phase.
Time Frame: Day 1 of Cycle 3, Day 1 of Cycle 5, and Day 22 of Cycle 6
Population: Participants who received at least 1 dose of study drug
Measure: Number; unit: Participants
Arm/Group | Dose Level 1: Ipilimumab, 3 mg/kg + Paclitaxel + Carboplatin | Dose Level 2: Ipilimumab, 10 mg/kg + Paclitaxel + Carboplatin
Number analyzed (Participants) | 8 | 7
Participants
  PR | 3 | 3
  Stable disease | 3 | 4

4. Secondary Outcome: Maximum Serum Concentration (Cmax) of Ipilimumab
Description: Cmax was recorded directly from experimental observations. Actual times were used for the analyses. Cmax measurements were performed during the 3rd cycle; at predose and at 1.5, 4 , 24 (Day 2), 48 (Day 3), 168 hrs (Day 8),and 336 (Day 15) hours postdose; during the 4th and subsequent cycle, predose ipilimumab; and off-treatment until progression of disease, toxicities requiring discontinuation, withdrawal of consent, or study closure.
Time Frame: During Cycle 3: predose and 1.5, 4, 24, 48, 168, and 336 hours postdose ipilimumab
Population: Participants who received at least 1 dose of ipilimumab
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Dose Level 1: Ipilimumab, 3 mg/kg + Paclitaxel + Carboplatin | Dose Level 2: Ipilimumab, 10 mg/kg + Paclitaxel + Carboplatin
Number analyzed (Participants) | 6 | 6
ug/mL | 72.8 (12) | 201 (21)

5. Secondary Outcome: Trough Observed Serum Concentration (Cmin) of Ipilimumab
Description: Cmin was recorded directly from experimental observations. Actual times were used for the analyses. Cmin measurements were performed during the 3rd cycle, at predose and at 1.5, 4 , 24 (Day 2), 48 (Day 3), 168 (Day 8), and 336 (Day 15) hours postdose; during the 4th and subsequent cycle, predose ipilimumab; and off-treatment until progression of disease, toxicities requiring discontinuation, withdrawal of consent; or study closure.
Time Frame: During Cycle 3: predose and 1.5, 4, 24, 48, 168, and 336 hours postdose ipilimumab
Population: Participants who received at least 1 dose of ipilimumab
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Dose Level 1: Ipilimumab, 3 mg/kg + Paclitaxel + Carboplatin | Dose Level 2: Ipilimumab, 10 mg/kg + Paclitaxel + Carboplatin
Number analyzed (Participants) | 6 | 6
ug/mL
  Day 22 | 11.06 (1.007) | 26.65 (4.599)
  Day 43 (n=3, 5) | 10.98 (4.773) | 26.68 (14.247)
  Day 64 (n=3, 3) | 13.90 (2.600) | 26.40 (7.904)

6. Secondary Outcome: Area Under the Concentration Curve From Time 0 to Day 21 (in 1 Interval Dosing) (AUC[0-21d]) for Ipilimumab
Description: The AUC(0-21d) was calculated using a mixture of log- and linear-trapezoidal summations. Using no weighting factor, the terminal log-liner phase of the concentration-time curve was determined by least-square linear regression of at least 3 data points. Individual patient pharmacokinetic (PK) parameter values were derived by noncompartmental methods using a validated PK analysis program. Actual times were used for the analyses. AUC(0-21d) measurements were performed during the 3rd cycle, at predose and at 1.5, 4 , 24 (Day 2), 48 (Day 3), 168 hrs (Day 8),and 336 (Day 15) hours postdose; during the 4th and subsequent cycle, predose ipilimumab; and off-treatment until progression of disease, toxicities requiring discontinuation, withdrawal of consent; or study closure.
Time Frame: During Cycle 3: predose and 1.5, 4, 24, 48, 168, and 336 hours postdose ipilimumab
Population: Participants who received at least 1 dose of ipilimumab
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug*h/mL
Arm/Group | Dose Level 1: Ipilimumab, 3 mg/kg + Paclitaxel + Carboplatin | Dose Level 2: Ipilimumab, 10 mg/kg + Paclitaxel + Carboplatin
Number analyzed (Participants) | 6 | 6
ug*h/mL | 12632 (12) | 36489 (21)

7. Secondary Outcome: Time of Maximum Observed Serum Concentration (Tmax)
Description: Tmax was recorded directly from experimental observations. Actual times were used for the analyses. Tmax measurements were performed during the 3rd cycle; at predose and at 1.5, 4 , 24 (Day 2), 48 (Day 3), 168 hrs (Day 8),and 336 (Day 15) hours postdose; during the 4th and subsequent cycle, predose ipilimumab; and off-treatment until progression of disease, toxicities requiring discontinuation, withdrawal of consent, or study closure.
Time Frame: During Cycle 3: predose and 1.5, 4, 24, 48, 168, and 336 hours postdose ipilimumab
Population: Participants who received at least 1 dose of ipilimumab
Measure: Median (Full Range); unit: Hours
Arm/Group | Dose Level 1: Ipilimumab, 3 mg/kg + Paclitaxel + Carboplatin | Dose Level 2: Ipilimumab, 10 mg/kg + Paclitaxel + Carboplatin
Number analyzed (Participants) | 6 | 6
Hours | 2.75 [1.37 to 4.08] | 3.98 [1.45 to 23.8]

8. Secondary Outcome: Serum Half-life (T-HALF) of Ipilimumab
Description: T-HALF was calculated as the ratio of ln(2) to elimination rate constant (K), where K was estimated as negative slope obtained by regression of the terminal log-linear portion of the serum concentration vs time profile following the ipilimumab dose on Day 1 of Cycle 3. Individual patient pharmacokinetic (PK) parameter values were derived by noncompartmental methods, using a validated PK analysis program. Actual times were used for the analyses. T-HALF measurements were performed during the 3rd cycle; at predose and at 1.5, 4 , 24 (Day 2), 48 (Day 3), 168 hrs (Day 8),and 336 (Day 15) hours postdose; during the 4th and subsequent cycle, predose ipilimumab; and off-treatment until progression of disease, toxicities requiring discontinuation, withdrawal of consent, or study closure.
Time Frame: During Cycle 3: predose and 1.5, 4, 24, 48, 168, and 336 hours postdose ipilimumab
Population: Participants who received at least 1 dose of ipilimumab
Measure: Mean (Standard Deviation); unit: Days
Groups:
- Dose Level 2: Ipilimumab, 10 mg/kg + Paclitaxel + Carboplatin: Participants received ipilimumab, 10 mg/kg, administered as a single dose IV over 90 minutes every 3 weeks, plus paclitaxel, 175 mg/m^2 , administered as a single dose IV over 3 hours every 3 weeks (up to 6 doses) and carboplatin, AUC=6, administered as a single dose IV over 30 -60 minutes every 3 weeks (up to 6 doses).
Arm/Group | Dose Level 1: Ipilimumab, 3 mg/kg + Paclitaxel + Carboplatin | Dose Level 2: Ipilimumab, 10 mg/kg + Paclitaxel + Carboplatin
Number analyzed (Participants) | 6 | 6
Days | 13.3 (3.64) | 11.3 (2.83)

ADVERSE EVENTS:
Arm/Group | Dose Level 1: Ipilimumab, 3 mg/kg + Paclitaxel + Carboplatin | Dose Level 2: Ipilimumab, 10 mg/kg + Paclitaxel + Carboplatin
Serious Adverse Events (participants affected / at risk) | 3/8 | 1/7
Other Adverse Events (participants affected / at risk) | 8/8 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Level 1: Ipilimumab, 3 mg/kg + Paclitaxel + Carboplatin (N=8) | Dose Level 2: Ipilimumab, 10 mg/kg + Paclitaxel + Carboplatin (N=7)
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoparathyroidism (Endocrine disorders) | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Level 1: Ipilimumab, 3 mg/kg + Paclitaxel + Carboplatin (N=8) | Dose Level 2: Ipilimumab, 10 mg/kg + Paclitaxel + Carboplatin (N=7)
Blood bilirubin increased (Investigations) | 0 | 1
Cheilitis (Gastrointestinal disorders) | 0 | 1
Cushingoid (Endocrine disorders) | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Eye inflammation (Eye disorders) | 1 | 0
Flushing (Vascular disorders) | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 4
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 2
Neutropenia (Blood and lymphatic system disorders) | 7 | 7
Stomatitis (Gastrointestinal disorders) | 2 | 1
Tinea pedis (Infections and infestations) | 1 | 0
Vitreous floaters (Eye disorders) | 1 | 0
Conjunctivitis (Eye disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1
Injection site erythema (General disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 5 | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 6 | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 6
Blood corticotrophin decreased (Investigations) | 0 | 1
Dysgeusia (Nervous system disorders) | 2 | 1
Eyelid oedema (Eye disorders) | 1 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 | 0
Weight decreased (Investigations) | 4 | 3
Weight increased (Investigations) | 0 | 1
Blood pressure decreased (Investigations) | 0 | 1
Blood sodium decreased (Investigations) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Gastritis (Gastrointestinal disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1
Hypothermia (General disorders) | 1 | 0
Injection site pain (General disorders) | 2 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 4
Respiratory tract haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 2
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Blood magnesium decreased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Dizziness postural (Nervous system disorders) | 1 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Lymphopenia (Blood and lymphatic system disorders) | 2 | 0
Metrorrhagia (Reproductive system and breast disorders) | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 7 | 6
Pyrexia (General disorders) | 3 | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 2
Somnolence (Nervous system disorders) | 1 | 0
Supraventricular extrasystoles (Cardiac disorders) | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Blood cortisol decreased (Investigations) | 0 | 1
Cystitis (Infections and infestations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 7 | 6
Dental caries (Gastrointestinal disorders) | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0
Tongue coated (Gastrointestinal disorders) | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1
Adrenal insufficiency (Endocrine disorders) | 1 | 0
Amylase increased (Investigations) | 2 | 2
Blood thyroid stimulating hormone decreased (Investigations) | 0 | 1
C-reactive protein increased (Investigations) | 2 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 2
Electrocardiogram QT prolonged (Investigations) | 4 | 2
Fatigue (General disorders) | 2 | 5
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1
Menorrhagia (Reproductive system and breast disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 6 | 5
Seasonal allergy (Immune system disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 4 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 2
Diverticulum (Gastrointestinal disorders) | 0 | 1
Duodenitis (Gastrointestinal disorders) | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 0 | 1
Gastric disorder (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Hypoaesthesia (Nervous system disorders) | 3 | 0
Insomnia (Psychiatric disorders) | 2 | 2
Leukopenia (Blood and lymphatic system disorders) | 4 | 2
Lipase increased (Investigations) | 0 | 1
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Retinal haemorrhage (Eye disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.